CLINICAL TRIAL: NCT01804621
Title: An RCT to Examine the Effects of Scanning; a Major Step on the Path Towards Population Intervention
Brief Title: RCT to Examine the Effects of Scanning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 811285; 3P20CA095856-07S1 (NIH)
Record Dates: First submitted 2013-02-25; First posted 2013-03-05 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2012-12

CONDITIONS: Cancer; Breast Cancer; Colorectal Cancer
Keywords: Exercise; Nutrition; Mammography; Colorectal screening
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Exercise (Experimental): Participant received health newsletter with targeted articles about exercise behavior.
  Interventions: Behavioral: Health Newsletter
- Fruit & Vegetable (Experimental): Participant received health newsletter with targeted articles about fruit & vegetable consumption.
  Interventions: Behavioral: Health Newsletter
- Colorectal Cancer Screening (Experimental): Participant received health newsletter with targeted articles about colorectal cancer screening.
  Interventions: Behavioral: Health Newsletter
- Mammography (Experimental): Participant received health newsletter with targeted articles about mammography screening.
  Interventions: Behavioral: Health Newsletter

INTERVENTIONS:
Behavioral: Health Newsletter — Participants received a health newsletter with articles about general health articles, as well as targeted health articles (differs by condition).

SUMMARY:
The purpose of the study is to implement a randomized control trial testing effects of information scanning on cancer prevention and screening behaviors in a population sample of 50-70 year olds. Participants will receive one of five versions of an e-newsletter once/month for 12 months and will be asked to complete baseline, mid-point, and end-of-project surveys.

ELIGIBILITY:
Inclusion Criteria:

* US adults, male or female, between 50 and 70 years of age.

Exclusion Criteria:

* Potential subjects will be excluded if they are not between the ages of 50 and 70

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15824 (Actual)
Dates: Start 2010-04; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Exercise Behavior | 12 months
  The Godin Scale was used to assess weekly exercise frequency and intensity
Fruit & Vegetable Consumption | 12 months
  Total daily servings of reported fruits and vegetables (maximum of 10) were calculated using a composite measure that summed separate responses for fruits and vegetables.
Mammography Screening Behavior | 12 months
  We used responses to two questions to create a dichotomous measure of whether or not female respondents (all aged 50 to 70) received a mammogram in the past year.
Colorectal cancer screening | 12 months
  A measure of up-to-date colorectal cancer screening status was assessed using individuals' self-reports of recency of colonoscopy (within 10 years), sigmoidoscopy (within five years), and/or fecal occult blood test (FOBT) within one year.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Hornik, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States